CLINICAL TRIAL: NCT01172093
Title: Prevalence and Recognition of Obstructive Sleep Apnea in Chinese With Type 2 Diabetes Mellitus
Brief Title: A Study on the Prevalence of Obstructive Sleep Apnea in Patients With Type II Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: The University of Hong Kong (Other)
Responsible Party: Professor Ip Sau Man Mary, The University of Hong Kong
Other Study IDs: UW07-060
Record Dates: First submitted 2010-07-27; First posted 2010-07-29 (Estimated); Last update posted 2010-07-29 (Estimated); Status verified 2010-07

CONDITIONS: Obstructive Sleep Apnea; Diabetes Mellitus
Keywords: obstructive sleep apnea; prevalence; diabetes mellitus; Chinese
MeSH Terms: conditions — Sleep Apnea, Obstructive; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Plasma and serum samples were collected from subjects for batch assays for further research purposes
Oversight: Data Monitoring Committee: Yes

SUMMARY:
OSA is prevalent among patients with type II DM

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) has been reported to be common (prevalence ranged from 23-86%) in previous studies involving Caucasian diabetic patients. The investigators aim at finding out the prevalence of OSA in Chinese diabetic patients and identify the clinical predictors associated with OSA.

Recruited subjects will undergo overnight polysomnography, anthropometric measurements, blood tests including glycosylated hemoglobin, renal function, glucose level, blood pressure measurement both during the clinic visit and after admission for in-laboratory sleep study.

ELIGIBILITY:
Inclusion Criteria:

* Patients, age 18 - 75, with type 2 diabetes mellitus, including those on diet, on oral-hypoglycaemic agents or on insulin
* Patients who are able to give written consent to undergo polysomnography

Exclusion Criteria:

* Patients who are unable or unwilling to give written consent to participate in the study
* Patients with unstable medical illness or poor functional performance
* Patients with recent myocardial infarction or hospital admission for congestive heart failure or cardiac arrhythmia in the past three months
* Patients on renal replacement therapy for diabetic nephropathy or chronic renal failure, or plan to start renal replacement therapy in the coming six months
* Patients suffered from recent stroke in the past six months or previous history of stroke with significant focal neurological deficit
* Patients with type I diabetes
* Pregnant lady or lactating women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All Chinese subjects with type 2 diabetes mellitus being followed up at the diabetic clinic of a University affiliated hospital
Sampling Method: Non-Probability Sample
Enrollment: 177 (Actual)
Dates: Start 2007-01; Primary Completion 2008-06 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
presence of OSA | measured at a single time point during the recruitment period(2007-08), by polysomnography
  The diagnosis of OSA will be confirmed with polysomnography

SECONDARY OUTCOMES:
severity of OSA | measured at a single time point during the recruitment period(2007-08), by polysomnography
  The severity of OSA will be assessed in terms of apnea hypopnea index, minimal oxygen saturation, duration of desaturation, arousal index during polysomnography
glycemic control | measured at a single time point, when the subjects were admitted for polysomnography (during 2007-08)
  by measuring glycosylated hemoglobin, blood glucose level

CONTACTS AND LOCATIONS:
Overall Officials: David CL Lam, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong

REFERENCES:
- [Background] Aronsohn RS, Whitmore H, Van Cauter E, Tasali E. Impact of untreated obstructive sleep apnea on glucose control in type 2 diabetes. Am J Respir Crit Care Med. 2010 Mar 1;181(5):507-13. doi: 10.1164/rccm.200909-1423OC. Epub 2009 Dec 17. PMID 20019340
- [Background] Elmasry A, Lindberg E, Berne C, Janson C, Gislason T, Awad Tageldin M, Boman G. Sleep-disordered breathing and glucose metabolism in hypertensive men: a population-based study. J Intern Med. 2001 Feb;249(2):153-61. doi: 10.1046/j.1365-2796.2001.00787.x. PMID 11240844
- [Background] Resnick HE, Redline S, Shahar E, Gilpin A, Newman A, Walter R, Ewy GA, Howard BV, Punjabi NM; Sleep Heart Health Study. Diabetes and sleep disturbances: findings from the Sleep Heart Health Study. Diabetes Care. 2003 Mar;26(3):702-9. doi: 10.2337/diacare.26.3.702. PMID 12610025
- [Background] West SD, Nicoll DJ, Stradling JR. Prevalence of obstructive sleep apnoea in men with type 2 diabetes. Thorax. 2006 Nov;61(11):945-50. doi: 10.1136/thx.2005.057745. Epub 2006 Aug 23. PMID 16928713
- [Background] Ronksley PE, Hemmelgarn BR, Heitman SJ, Hanly PJ, Faris PD, Quan H, Tsai WH. Obstructive sleep apnoea is associated with diabetes in sleepy subjects. Thorax. 2009 Oct;64(10):834-9. doi: 10.1136/thx.2009.115105. Epub 2009 Aug 12. PMID 19679579
- [Background] Foster GD, Sanders MH, Millman R, Zammit G, Borradaile KE, Newman AB, Wadden TA, Kelley D, Wing RR, Sunyer FX, Darcey V, Kuna ST; Sleep AHEAD Research Group. Obstructive sleep apnea among obese patients with type 2 diabetes. Diabetes Care. 2009 Jun;32(6):1017-9. doi: 10.2337/dc08-1776. Epub 2009 Mar 11. PMID 19279303
- [Derived] Lam DC, Lui MM, Lam JC, Ong LH, Lam KS, Ip MS. Prevalence and recognition of obstructive sleep apnea in Chinese patients with type 2 diabetes mellitus. Chest. 2010 Nov;138(5):1101-7. doi: 10.1378/chest.10-0596. Epub 2010 Aug 12. PMID 20705796